CLINICAL TRIAL: NCT03173521
Title: A Phase I/II Open Label, Dose Escalation, Safety Study in Subjects With Mucopolysaccharidosis Type VI (MPS VI) Using Adeno-Associated Viral Vector 8 to Deliver the Human ARSB Gene to Liver
Brief Title: Gene Therapy in Patients With Mucopolysaccharidosis Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Telethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIGEM1-MPS VI
Record Dates: First submitted 2017-04-12; First posted 2017-06-02 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Mucopolysaccharidosis Type VI
Keywords: MPSVI
MeSH Terms: conditions — Mucopolysaccharidosis VI

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label (Experimental): Adeno-associated viral vector serotype 8 with liver-specific thyroxine-binding globulin (TBG) promoter driving the expression of the human ARSB gene diluted in its final formulation medium [Drug product (DP) diluted in 0.9% saline solution and 0.25% of human serum albumin].
  Four dose levels are available:
  * 'Starting dose' is 6x1011 gc of vector per kg of body weight.
  * 'High dose' is 2x1012 gc of vector per kg of body weight.
  * 'Very high dose' is 6x1012 gc of vector per kg of body weight.
  * 'Low dose' is 2x1011 gc of vector per kg of body weight. Intermediate doses are also possible. The administration of the IMP will be performed into a peripheral vein (e.g. median cubital vein) over 2-4 hours using an infusion pump. The IMP final volume to be injected is calculated based on the patient's weight (determined on the day of hospital admission), as 3 mL/kg.
  Interventions: Biological: AAV2/8.TBG.hARSB

INTERVENTIONS:
Biological: AAV2/8.TBG.hARSB — Adeno-associated viral vector serotype 8 with liver-specific thyroxinebinding globulin (TBG) promoter driving the expression of the human ARSB gene. Four dose levels are available:
  * Starting dose is 6x1011 gc of vector per kg of body weight;
  * High dose is 2x1012 gc of vector per kg of body weight and will be administered after at least two subjects at the starting dose have experienced no DLT;
  * Very high dose is 6x1012 vector per kg of body weight and will be administered after three subjects at the high dose have experienced no DLT;
  * Low dose is 2x1011 gc of vector per kg of body weight. Intermediate doses are also possible. The administration of the IMP will be performed into a peripheral vein. The IMP final volume to be injected is calculated based on the patient's weight (determined on the day of hospital admission), as 3 mL/kg.

SUMMARY:
This study investigated the safety and efficacy of gene therapy approaches for Mucopolysaccharidosis type VI disease caused by the deficiency of arylsulfatase B (ARSB) enzyme. The aim of the study is to evaluate the safety and efficacy of the treatment.

DETAILED DESCRIPTION:
Mucopolysaccharidosis type VI disease is involved in Lysosomal Storage Disorder. The MPS VI disease is characterized by growth retardation, corneal clouding, cardiac valve disease, organomegaly, skeletal dysplasia, without central nervous system involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Documented biochemical and molecular diagnosis of MPS VI. Testing for homozygous or compound heterozygous disease-causing mutations of the ARSB gene must have been performed by an accredited laboratory.
2. Subjects must be of 4 years of age or older.
3. Subjects should have received ERT for at least 12 months before enrolment and should continue to receive ERT until 7-14 days before IMP administration.
4. Documented informed consent; willingness to adhere to protocol and to participate to long-term follow-up, as evidenced by written informed consent.

Exclusion Criteria:

1. Subjects unable or unwilling to meet requirements of the study.
2. Participation in a clinical study with an investigational drug in the 6 months prior to enrolment in this trial.
3. Subjects unable to perform the 6MWT.
4. History of severe anaphylactoid reaction to Naglazyme in subjects receiving ERT that could affect the safety (severe reaction is meant to be a respiratory impairment event that is life-threatening).
5. Presence of tracheostomy or need of ventilatory assistance.
6. Subjects with evidence of progressive myelomalacia that is considered severe enough to require neck surgery in the first six months after enrolment.
7. Values of AST or ALT above the upper limit of normal range at baseline 2 (at -5days) evaluations.
8. Co-existence of chronic diseases or clinically relevant abnormal baseline laboratory values; infections with hepatitis B, C, or HIV (Baseline 1).
9. Systemic corticosteroid therapy or other immunosuppressive/immunomodulating drugs within 2 months prior to IMP administration.
10. Female individuals of childbearing age who are pregnant or nursing or unwilling to use effective contraception for at least one year post-IMP administration.
11. Fertile male individuals who are unwilling to use male barrier contraceptives such as condom.
12. Any other condition that would not allow the subject to complete follow-up examinations during the course of the study and that, in the opinion of the Investigator, would make the subject unsuitable for the study.
13. Presence of serum NAB to AAV8 above the limit of detection of the assay (Screening and Baseline 1).
14. Presence of serum antibodies anti-ARSB above the upper limit of detection of the assay (antibodies anti-ARSB level >31250 or declared positive at the value of serum dilution 1.10 according to the performed assay) at Screening and Baseline 1.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the IMP administration | From GT up to 5 years post IMP administration at the following visits: days 1,2,3; weeks 2,3,6,7,8,9,10,11,12,13,14; months 4,9,12; years 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5.
  Overall safety and tolerability will be determined through monitoring of adverse events, laboratory and clinical investigations and imaging studies (for example complete physical examination with vital signs recording, liver ultrasound, measurement of transaminases, thyroids hormones, creatinine, albumin, total proteins in blood and urine, and urea, C3 and C4 in blood).
Primary efficacy outcome - Urinary GAG levels | From GT up to 5 years post IMP administration at the following visits: days 1,2,3; months 4,9,12,15; years 1.5,1.75, 2, 2.5, 3, 4, 5.
  To determine the efficacy of gene therapy, post-injection urinary GAG excretion levels will be compared to the average of pre-injection urinary GAG determined at baseline 1 and at visit 1.

SECONDARY OUTCOMES:
Secondary efficacy outcome - endurance | From GT up to 5 years post IMP administration at the following visits: months 4,9,12; years 1.5, 2, 2.5, 3.
  Endurance as measured by 6-minute walk test (6MWT) in walking subjects, 3-minute stair climb test (3MSCT) in walking subjects.
Secondary efficacy outcome - lung volumes | From GT up to 5 years post IMP administration at the following visits: months 4,9,12; years 1.5, 2, 2.5, 3.
  Forced vital capacity (FVC), and forced expiratory volume at 1 second (FEV1) in cooperative subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Brunetti-Pierri, Principal Investigator — Department of Translational Medicine (DISMET) of "Federico II" University, Naples
Locations (2):
- Department of Translational Medicine (DISMET) of "Federico II" University, Naples, Naples, Italy
- Children's Hospital Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Rossi A, Romano R, Fecarotta S, Dell'Anno M, Pecorella V, Passeggio R, Zancan S, Parenti G, Santamaria F, Borgia F, Deodato F, Funghini S, Rupar CA, Prasad C, O'Callaghan M, Mitchell JJ, Valsecchi MG, la Marca G, Galimberti S, Auricchio A, Brunetti-Pierri N. Multi-year enzyme expression in patients with mucopolysaccharidosis type VI after liver-directed gene therapy. Med. 2025 Apr 11;6(4):100544. doi: 10.1016/j.medj.2024.10.021. Epub 2024 Nov 14. PMID 39547230
- [Derived] Brunetti-Pierri N, Ferla R, Ginocchio VM, Rossi A, Fecarotta S, Romano R, Parenti G, Yildiz Y, Zancan S, Pecorella V, Dell'Anno M, Graziano M, Alliegro M, Andria G, Santamaria F, Brunetti-Pierri R, Simonelli F, Nigro V, Vargas M, Servillo G, Borgia F, Soscia E, Gargaro M, Funghini S, Tedesco N, Le Brun PR, Rupar CA, Prasad C, O'Callaghan M, Mitchell JJ, Danos O, Marteau JB, Galimberti S, Valsecchi MG, Veron P, Mingozzi F, Fallarino F, la Marca G, Sivri HS, Auricchio A. Liver-Directed Adeno-Associated Virus-Mediated Gene Therapy for Mucopolysaccharidosis Type VI. NEJM Evid. 2022 Jul;1(7):EVIDoa2200052. doi: 10.1056/EVIDoa2200052. Epub 2022 Jun 6. PMID 38319253